CLINICAL TRIAL: NCT02551549
Title: A Phase 1, Randomized, Double-Blind, Multiple-Dose, Dose-Escalation Study to Determine the Safety, Tolerability, and Pharmacokinetics of CD101 Injection in Healthy Subjects
Brief Title: An Ascending Multiple Dose Study of CD101 IV in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cidara Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CD101.IV.1.02
Record Dates: First submitted 2015-09-14; First posted 2015-09-16 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Healthy
Keywords: Subjects
MeSH Terms: interventions — echinocandin CD101 IV

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CD101 IV (Experimental): multiple ascending dose intravenous infusion
  Interventions: Drug: CD101 IV
- Placebo (Placebo Comparator): normal saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CD101 IV — antifungal
  Arms: CD101 IV
Drug: Placebo — Normal saline
  Arms: Placebo

SUMMARY:
A multiple ascending dose study to evaluate the safety, tolerability, and pharmacokinetics of CD101 Injection in Healthy Subjects.

DETAILED DESCRIPTION:
This is a Phase 1, single-center, prospective, randomized, double-blind study of multiple ascending doses (MAD) of CD101 Injection administered IV to healthy adult subjects. In this study, subjects in 3 cohorts of 8 subjects each will be randomized to receive multiple IV doses of CD101 Injection or placebo infusions. Dose levels of CD101 Injection to be assessed will follow an ascending multiple-dose regimen.

ELIGIBILITY:
Inclusion Criteria:

* Men must be surgically sterilized or using contraception,
* No significant findings on physical exam, ECG, clinical laboratory tests,
* Body mass index (BMI) between 18.5 and 32.0 kg/m2, inclusive
* Must provide written informed consent

Exclusion Criteria:

* Females of child bearing potential
* Signs and or symptoms of acute illness or chronic disease
* Use of prescription medications within 28 days
* Use of OTC, supplements, and herbals within 14 days
* Current smoker
* Previous participation in a clinical study within 28 days

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-09; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Safety as assessed by the number of subjects with clinically significant adverse events | Up to 2 weeks following last dose of study drug
  Number of subjects with clinically significant adverse events (AEs)

SECONDARY OUTCOMES:
Peak plasma concentration (Cmax) | Up to 2 weeks following last dose of study drug
Time to reach peak plasma concentration (Tmax) | Up to 2 weeks following last dose of study drug
Area under the concentration time curve (AUC) | Up to 2 weeks following last dose of study drug
The volume of plasma cleared of the drug per unit time (CL) | Up to 2 weeks following last dose of study drug
Apparent volume in which the drug is distributed (Vz) | Up to 2 weeks following last dose of study drug
The rate at which a drug is removed from the body (^z), | Up to 2 weeks following last dose of study drug
Terminal half-life (t1/2) | Up to 2 weeks following last dose of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Armas, MD, Principal Investigator — Celerion
Locations (1):
- Celerion Inc, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided